CLINICAL TRIAL: NCT00060489
Title: Safety and Efficacy Trial of the Use of Quetiapine Fumarate (SEROQUEL®) in the Treatment of Patients With Bipolar Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Purpose: Treatment
Other Study IDs: 5077US/0049
Record Dates: First submitted 2003-05-06; First posted 2003-05-08 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2011-01

CONDITIONS: Bipolar Disorder; Depression, Bipolar
Keywords: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — Quetiapine Fumarate; Tablets

INTERVENTIONS:
Drug: SEROQUEL (quetiapine fumarate) Tablets

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of quetiapine in the treatment of a major depressive episode in patients with bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent;
* Bipolar disorder with most recent episode depressed;
* Outpatient status

Exclusion Criteria:

* Patients with a current Axis I disorder other than bipolar disorder within 6 months of screening;
* Patients whose current episode of depression exceeds 12 months or is less than 4 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-09; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Birmingham, Alabama
  - Beverly Hills, California
  - La Mesa, California
  - San Diego, California
  - Jacksonville, Florida
  - Orlando, Florida
  - West Palm Beach, Florida
  - Winter Park, Florida
  - Atlanta, Georgia
  - Smyrna, Georgia
  - Oak Brook, Illinois
  - Shreveport, Louisiana
  - Clementon, New Jersey
  - Moorestown, New Jersey
  - New York, New York
  - Staten Island, New York
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Columbia, South Carolina
  - Memphis, Tennessee
  - Austin, Texas
  - Salt Lake City, Utah
  - Falls Church, Virginia
  - Bellevue, Washington
  - Kirkland, Washington

REFERENCES:
- [Derived] Lydiard RB, Culpepper L, Schioler H, Gustafsson U, Paulsson B. Quetiapine monotherapy as treatment for anxiety symptoms in patients with bipolar depression: a pooled analysis of results from 2 double-blind, randomized, placebo-controlled studies. Prim Care Companion J Clin Psychiatry. 2009;11(5):215-25. doi: 10.4088/PCC.08m00659. PMID 19956459